CLINICAL TRIAL: NCT03794232
Title: Study on the Mechanisms of Soluble Dietary Fiber Extracted From Jerusalem Artichoke in the Treatment of Pre-type 2 Diabetes
Brief Title: Effect of Inulin-type Fructose Extracted From Jerusalem Artichoke on Improving Prediabetic State of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inuling (Bei Jing) Science and Technology Co. Ltd (Industry)
Collaborators: Peking Union Medical College Hospital (Other); Proswell Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-749
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-11

CONDITIONS: Prediabetes
Keywords: Inulin; Soluble dietary fiber; Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): NIUCHANG（Soluble dietary fiber + prebiotics）：Oral, 1 bag (15g) once a day, taking 24 weeks
  Interventions: Dietary Supplement: NIUCHANG
- Control group (Placebo Comparator): Placebo（inactive drug ingredient）：Oral, 1 bag (15g) once a day, taking 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NIUCHANG
  Arms: Test group
Dietary Supplement: Placebo
  Arms: Control group

SUMMARY:
The trial was a multicenter, randomized, double-blind, placebo-controlled, parallel-controlled, exploratory clinical study.Through the intervention of soluble dietary fiber in the pre-type 2 diabetic population, the change of blood glucose spectrum before and after intervention can show the effect of this intervention on the outcome, and further elucidate the effect of soluble dietary fiber intervention on the level of insulin resistance and its effect on outcome. Helps to prevent the more scientific and effective prevention of type 2 diabetes from pre-diabetes.

Subjects who met the criteria were randomly divided into the experimental group and the control group, after 24 weeks of intervention, the incidence of blood sugar reversion to normal was main observed.The main purpose of this study was to investigate the effect of soluble dietary fiber treatment regimens on the conversion rate of pre-type 2 diabetes (converted to normal blood glucose, type 2 diabetes, or stable in the stage of impaired glucose tolerance). The secondary objective was to study the improvement of insulin resistance and changes in intestinal flora after intervention.

DETAILED DESCRIPTION:
The soluble dietary fiber (NIUCHANG®) and placebo used in the trial were exclusively produced by Inuling (Beijing) Technology Co., Ltd. and provided free of charge. During the treatment period, the treatment group was given oral "NIUCHANG®" (once 15g,once a day)and the control group was given oral placebo (once15 g, once a day) for 24 weeks.

The test was performed for 12 weeks as a course of treatment。At the end of one course of treatment, if the glucose tolerance was changed to normal or the blood glucose was stable in the pre-diabetes phase, the original dose was maintained and continued for 12 weeks. At 24 weeks, patients with normal blood glucose and glucose tolerance tests were followed up for 48 weeks. At the end of one course of treatment, if the blood glucose progresses to the stage of diabetes, the test is withdrawn and treated according to clinical routine.

ELIGIBILITY:
Inclusion Criteria:

The following various situations need to be met at the same time in order to be selected:

* According to the diagnostic criteria for impaired glucose tolerance in the WHO Diabetes Diagnosis and Classification Standard in 1999: fasting blood glucose ≥6.1mmol/L and <7.0mmol/L, blood glucose 2 hours after oral administration of 75g glucose ≥7.8mmol/L and < 11.1mmol/L;
* BMI：20kg/㎡ ≤ BMI ≤ 35kg/㎡；
* Age ≥ 18 and ≤ 70 years old, gender is not limited;
* Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

Any of the following circumstances should be excluded and cannot be selected:

* Acute cardiovascular and cerebrovascular events or myocardial infarction within 6 months;
* Laboratory examination: liver function AST or ALT ≥ 2.5 × ULN; renal function Cr > 1.2 × ULN;
* Those with severe gastrointestinal diseases, such as active peptic ulcer, intestinal obstruction, etc.; those who have changed the history of normal structure of the gastrointestinal tract;
* Hypertensive patients with poor blood pressure control (blood pressure SBP ≥ 160 mmHg and / or DBP ≥ 100 mmHg);
* Those with severe blood system diseases;
* Those with other endocrine system diseases, such as hyperthyroidism or hypercortisolism;
* Those who have a stress state or have secondary blood glucose elevation factors (such as those who take glucocorticoids);
* Women who are pregnant or breast-feeding, who are planning to be pregnant or who are not willing to contraception during the study;
* Drug or other drug abusers;
* Those who may be allergic to the test drug;
* Those who have participated in other drug trials within 3 months;
* Those who are unable to cooperate with mental illness;
* Other circumstances The investigator believes that it is not suitable for the group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence of blood sugar reversal to normal after intervention | Day 0, Week 24
  Through the intervention of soluble dietary fiber in the pre-diabetic population, the change of blood glucose spectrum before and after intervention can show the effect of this intervention on the outcome, and further elucidate the effect of soluble dietary fiber intervention on the level of insulin resistance and its effect on outcome.

SECONDARY OUTCOMES:
Changes in insulin resistance index | Day 0, Week 24
  the incidence of blood sugar reversion to normal was main observed
Changes in intestinal flora | Day 0, Week1，Week4，Week12，Week 24
  If the subject has had diarrhea or taking antibiotics 2 days before and after the fecal specimen should be taken, wait for the stagnation for 1 week before taking the stool specimen to reduce the interference of external factors.
Incidence of blood glucose stabilization in pre-diabetes after intervention | Day 0, Week12，Week 24
  blood glucose becomes stable
Incidence of blood glucose progression to diabetes after intervention | Day 0, Week12，Week 24
  reduce incidence of blood glucose progression
Hemoglobin A1C、Glycated Albumin | Day 0, Week 24
  Changes of Hemoglobin A1C and Glycated Albumin.
The levels of serum insulin | Day 0, Week 24
  Insulin levels were measured on an empty stomach, 30 minutes, 60 minutes and 120 minutes after oral administration of 75 g of glucose.
The levels of serum C-peptid | Day 0, Week 24
  C-peptide levels were measured on an empty stomach, 30 minutes, 60 minutes and 120 minutes after oral administration of 75 g of glucose.
Body weight | Day 0, Week12，Week 24
  Changes of body weight.